CLINICAL TRIAL: NCT01432145
Title: Phase II Clinical Trial Of 6-Mercaptopurine (6MP) and Low-Dose Methotrexate In Patients With Known BRCA Defective Tumours
Brief Title: A Clinical Trial in Patients With Breast Cancer Susceptibility Gene (BRCA) Defective Tumours
Acronym: 6MP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCTO_016
Record Dates: First submitted 2011-08-10; First posted 2011-09-12 (Estimated); Results first posted 2019-05-17 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2018-06

CONDITIONS: Breast Cancer; Ovarian Cancer
Keywords: BRCA defective
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms | interventions — Mercaptopurine; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 6MP/MTX (Experimental): 6-Mercaptopurine 55mg/m2 per day, and methotrexate 15mg/m2 per week
  Interventions: Drug: 6-Mercaptopurine; Drug: Methotrexate

INTERVENTIONS:
Drug: 6-Mercaptopurine — 6-Mercaptopurine (6MP) 55mg/m2 body surface area, administered orally (PO) once a day (od) in the morning 1 hour after eating, on a continuous schedule. One cycle is 28 days. Treatment is given continuously until disease progression.
  Other Names: 6MP
Drug: Methotrexate — Methotrexate (MTX) 15 mg/m2 taken orally, once a week, in the morning. One cycle is 28 days. Treatment is given continuously until disease progression.
  Other Names: MTX

SUMMARY:
This study will evaluate the efficacy and safety of 6-mercaptopurine (6MP) in combination with methotrexate (MTX) in patients with breast or ovarian cancer who are known to have a BRCA (breast cancer gene) mutation.

DETAILED DESCRIPTION:
This study will evaluate the efficacy and safety of 6-mercaptopurine (6MP) in combination with methotrexate (MTX) in patients with breast or ovarian cancer who are known to have a BRCA (breast cancer gene) mutation. 6MP is used instead of thioguanine(6TG) as it is converted to the same cytotoxic moiety as 6TG, ie. thioguanine nucleotides, but with reduced toxic effects. Low dose methotrexate is used in combination with 6MP as it promotes the formation of thioguanine nucleotides.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with proven BRCA1 or BRCA2 mutations and after appropriate exposure to standard treatment, as defined by:

   Breast Cancer
   * Patients with initially histologically or cytologically proven locally advanced or metastatic breast cancer who may have received up to 3 previous lines of chemotherapy in the locally advanced or metastatic breast cancer setting.
   * Patients must have previously had a taxane and an anthracycline in either the adjuvant or metastatic setting, provided that these were not contraindicated.
   * Patients with hormone responsive disease should have had at least 1 line of hormone therapy for metastatic disease.
   * Prior treatment with a poly-Adenosine diphosphate (ADP) ribose polymerase (PARP) inhibitor is permissible.

   OR Ovarian Cancer
   * Patients with initially histologically or cytologically proven ovarian cancer.
   * Patients must have disease that is platinum resistant or in whom further platinum based therapy is inappropriate.
   * Prior treatment with a PARP inhibitor is permissible.
2. Patients must have measurable disease on computerized tomography (CT) or Magnetic resonance imaging (MRI) scan as defined by Response Evaluation Criteria In Solid Tumors (RECIST) criteria.
3. Age ≥18 years.
4. Eastern Cooperative Oncology Group (ECOG) performance score of 0-2.
5. Life expectancy >12 weeks.
6. Written informed consent.
7. Patient willing and able to comply with all protocol requirements.
8. No prior anti-cancer treatment in previous 4 weeks, other than palliative radiotherapy (RT).
9. Haematological and biochemical indices within the ranges shown below.

   * Laboratory Test Value required
   * Haemoglobin (Hb) > 10g/dL
   * White Blood Count (WBC) > 3x109/L
   * Platelet count > 100,000/μL
   * Absolute Neutrophil count > 1.5x109/L;
   * Serum bilirubin ≤ 2 x Upper limit normal (ULN)
   * Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase (SGOT)) and alanine aminotransferase (ALT) or ALT ≤ 5 x ULN (liver metastasis)
   * or ≤ 3 x ULN (no liver metastasis)
   * Alkaline phosphatase ≤ 5 x ULN
   * Serum creatinine ≤ 1.5 x ULN
10. Ascites and pleural effusions must be drained prior to therapy.

Exclusion Criteria:

1. Patients with any of the following contra-indications to thiopurines (6MP or 6TG) or methotrexate:

   * family history of severe liver failure;
   * alcoholism;
   * porphyria;
   * diffuse infiltrative pulmonary or pericardial disease;
   * known hypersensitivity to either trial agent.
2. Patients found to have a Low/Low genotype on thiopurine methyltransferase (TPMT) testing will be excluded.
3. Pregnant or breast-feeding women or women of childbearing potential unless highly effective methods of contraception are used.
4. Other active malignancy, with the exception of adequately treated in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin.
5. Patients known or tested to be serologically positive for Hepatitis B, Hepatitis C or human immunodeficiency virus (HIV).
6. Patients with active central nervous system (CNS) lesions are excluded (i.e., those with radiographically unstable, symptomatic lesions). However, patients treated with stereotactic therapy or surgery and/or whole brain radiotherapy are eligible if the patient remains without evidence of disease progression in brain ≥ 3 months prior to registration date . They must also be off corticosteroid therapy for ≥ 3 weeks prior to registration date.
7. Patients who have received anticancer agent(s) or an investigational agent within 28 days prior to study drug administration.
8. Subjects who have not recovered to within one grade level (not to exceed grade 2) of their baseline following a significant adverse event or toxicity attributed to previous anticancer treatment are excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2011-05; Primary Completion 2014-12 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shibani Nicum, Principal Investigator — University of Oxford
Locations (1):
- Churchill Hospital, Oxford, United Kingdom

REFERENCES:
- [Derived] Roberts C, Strauss VY, Kopijasz S, Gourley C, Hall M, Montes A, Abraham J, Clamp A, Kennedy R, Banerjee S, Folkes LK, Stratford M, Nicum S. Results of a phase II clinical trial of 6-mercaptopurine (6MP) and methotrexate in patients with BRCA-defective tumours. Br J Cancer. 2020 Feb;122(4):483-490. doi: 10.1038/s41416-019-0674-4. Epub 2019 Dec 9. PMID 31813938
- [Derived] Nicum S, Roberts C, Boyle L, Kopijasz S, Gourley C, Hall M, Montes A, Poole C, Collins L, Schuh A, Dutton SJ; 6MP Collaborative Group. A phase II clinical trial of 6-mercaptopurine (6MP) and methotrexate in patients with BRCA defective tumours: a study protocol. BMC Cancer. 2014 Dec 19;14:983. doi: 10.1186/1471-2407-14-983. PMID 25526776

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 74 patients were consented and registered from 14 sites between May 2011 and October 2014, and 67 of these registered patients were found to be evaluable. This is larger than the planned sample size of 65 patients, to compensate for unevaluable patients.
Pre-assignment Details: No wash out or run-in periods. No enrolled participants were excluded from the study before assignment.
Groups:
- 6MP/MTX: 6-Mercaptopurine: The dose of 6MP will be 75mg/m2 body surface area, administered orally (PO) once a day (od) in the morning 1 hour after eating, on a continuous schedule. Tablets should be taken at roughly the same time each day. One cycle is 28 days. Treatment is given continuously until disease progression.
  Methotrexate: Methotrexate (20 mg/m2) will be taken orally, once a week, in the morning. One cycle is 28 days. Treatment is given continuously until disease progression.
  Update: These original doses were reduced following an Urgent Safety Measure in August 2012 due to a large proportion of patients requiring a dose reduction or treatment delay due to incidences of myelo-suppression.
  The reduced doses were 55mg/m2 of 6MP orally once a day, and 15mg/m2 of Methotrexate orally once a week.
Period: Overall Study
Arm/Group | 6MP/MTX
Started | 74 (Corrected from 75. 75 was entered in error)
Completed | 67
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | 6MP/MTX
Number analyzed (Participants) | 67
Age, Continuous [Mean (Full Range); unit: years] | 55.9 [32 to 80]
Age, Customized [Count of Participants; unit: Participants]
  Age categorical: 18-64 years | 54
  Age categorical: 65-84 years | 13
  Age categorical: 85 years and over | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 67
Breast Cancer gene (BRCA) Status [Count of Participants; unit: Participants]
  BRCA 1 | 40
  BRCA 2 | 27
Prior poly-Adenosine diphosphate (ADP) ribose polymerase (PARP) treatment [Count of Participants; unit: Participants]
  Yes | 26
  No | 41
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG performance status is a scale used to assess how a patient's disease is progressing, assess how the disease affects the daily living abilities of the patient, and determine appropriate treatment and prognosis.
  Grade 0: fully active. Grade 1: restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature Grade 2: up and about more than 50% of waking hours Grade 3: confined to bed or chair more than 50% of waking hours Grade 4: completely disabled Grade 5: dead
  Participants
    PS 0 | 27
    PS 1 | 36
    PS 2 | 4
Albumin levels [Mean (Full Range); unit: g/dl] | 39.8 [28 to 49]
Thiopurine methyltransferase (TPMT) [Mean (Full Range); unit: mU/L] | 88.3 [43 to 160]

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate to 6-mercaptopurine and Methotrexate (6MP/MTX) in This Patient Population.
Description: 1st stage: If less than 3/30 evaluable patients respond at 8 weeks the trial will be stopped for futility. If 3 or more out of 30 evaluable patients respond then a further 35 patients will be recruited (2nd stage) - this was met.
  The proportion of patients responding to treatment (complete response, partial response or stable disease) at the second stage will be presented per Response Evaluation Criteria In Solid Tumours (RECIST) criteria version 1.1 measured radiologically with computerised tomography (CT) and/or magnetic resonance imaging (MRI); the same method is used at baseline and at follow-up: Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. Patients who yield progressive disease (PD) are classed as non-responders.
Time Frame: 8 weeks after start of treatment
Population: Evaluable patients are those patients who complete at least 4 out of 8 weeks of trial medication and are assessed for response as per RECIST v1.1 at 8 weeks. Patient who stop trial medication early due to disease progression are also fully evaluable as they have reached an end point.
Measure: Count of Participants; unit: Participants
Groups:
- 6-Mercaptopurine and Methotrexate (6MP/MTX): 6-Mercaptopurine: 6MP 75mg/m2 body surface area, administered orally (PO) once a day (od) in the morning 1 hour after eating, on a continuous schedule. One cycle is 28 days. Treatment is given continuously until disease progression.
  Methotrexate: Methotrexate 20mg/m2 will be taken orally, once a week, in the morning. One cycle is 28 days. Treatment is given continuously until disease progression.
  Update: These original doses were reduced following an Urgent Safety Measure in August 2012 due to a large proportion of patients requiring a dose reduction or treatment delay due to incidences of myelo-suppression.
  The reduced doses were 55mg/m2 of 6MP orally once a day, and 15mg/m2 of Methotrexate orally once a week.
Arm/Group | 6-Mercaptopurine and Methotrexate (6MP/MTX)
Number analyzed (Participants) | 67
Participants | 22

2. Secondary Outcome: Quality of Life - EuroQol Group, Five Dimensions, Three-level (EQ-5D-3L) Standardized Instrument for Measuring Generic Health Status
Description: Evaluated using the EQ-5D-3L questionnaire at baseline, 3 and 6 months, and at the end of treatment or 12 months, as well as using the ECOG performance status measure after each cycle
Time Frame: At the end of treatment or 12 months
Population: Quality of life could not be analysed due to the low questionnaire completion rate; only two patients (3%) completed the baseline and 12 month follow up QoL questionnaires, , but data could not be reported in the Outcome Measure due to confidentiality issues.
Arm/Group | 6-Mercaptopurine and Methotrexate (6MP/MTX)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From start of treatment until end of follow-up, up to 2 years.
Description: For Adverse Events (AEs), Grade 3 and 4 AEs and Grade 2 Adverse Drug Reactions (ADRs) were collected.
Groups:
- 6MP/MTX: 6-Mercaptopurine: The dose of 6MP will be 75mg/m2 body surface area, administered orally (PO) once a day (od) in the morning 1 hour after eating, on a continuous schedule. Tablets should be taken at roughly the same time each day. One cycle is 28 days. Treatment is given continuously (see table below) until disease progression.
  Methotrexate: Methotrexate (20 mg/m2) will be taken orally, once a week, in the morning. One cycle is 28 days. Treatment is given continuously (see table below) until disease progression.
Arm/Group | 6MP/MTX
All-Cause Mortality (participants affected / at risk) | 52/67
Serious Adverse Events (participants affected / at risk) | 33/67
Other Adverse Events (participants affected / at risk) | 46/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 6MP/MTX (N=67)
Thromboembolic event (Vascular disorders) | 3
Neutrophil count decreased (Investigations) | 6
Palpitations (Cardiac disorders) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Ataxia (Nervous system disorders) | 1
Fever (General disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 5
Ascites (Gastrointestinal disorders) | 1
Colonic obstruction (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Urinary tract obstruction (Renal and urinary disorders) | 1
Obstruction (Hepatobiliary disorders) | 1 — Blocked biliary stent
Female genital tract fistula (Reproductive system and breast disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Anorectal infection (Infections and infestations) | 1
Infection (Infections and infestations) | 1 — Temperature of 39.9 degrees celsius and feeling generally unwell. Infective process suspected but throat swab, urine, stool samples, blood cultures all negative. Treated with IV antibiotics. Source of infection not identified.
Lung infection (Infections and infestations) | 3
Sepsis (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 6MP/MTX (N=67)
Neutrophil count decreased (Investigations) | 24 (41)
Platelet count decreased (Investigations) | 5 (8)
White blood cell count decreased (Investigations) | 15 (21)
Anaemia (Blood and lymphatic system disorders) | 22 (27)
Fatigue (General disorders) | 19 (24)
Ascites (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 12 (15)
Vomiting (Gastrointestinal disorders) | 9 (11)
Abdominal pain (Hepatobiliary disorders) | 8 (9)
Urinary tract infection (Infections and infestations) | 3 (3)
Alanine Aminotransferase Increased (Investigations) | 4 (9)
Anorexia (Metabolism and nutrition disorders) | 3 (5)
Blood bilirubin increased (Investigations) | 4 (6)
Diarrhoea (Gastrointestinal disorders) | 3 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
GGT increased (Investigations) | 3 (5)
Headache (Nervous system disorders) | 3 (3)
Mucositis Oral (Gastrointestinal disorders) | 6 (6)

LIMITATIONS AND CAVEATS:
Quality of life, a secondary endpoint, could not be analysed due to the low questionnaire completion rate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI Publication needs to be after the first study multip-centre publication and make reference to it.